CLINICAL TRIAL: NCT04674449
Title: International Study of Coronary Microvascular Angina (iCorMicA): a Randomised, Controlled, Multicentre Trial and Registry
Brief Title: iCorMicA - Stratified Medicine in Angina
Acronym: iCorMicA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: GN19CA435
Record Dates: First submitted 2020-06-24; First posted 2020-12-19 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Microvascular Angina; Angina, Stable; Ischemia With No Obstructive Coronary Arteries (INOCA); Coronary Microvascular Dysfunction (CMD); Ischaemic Heart Disease; Non-Obstructive Coronary Atherosclerosis; Coronary Artery Disease; Vasospastic Angina; Coronary; Ischemic; Angina Attacks
Keywords: angina; microvascular angina; ischaemia with no obstructive coronary artery disease (INOCA); stratified medicine; clinical trial; outcomes research; prognosis; health economics
MeSH Terms: conditions — Microvascular Angina; Angina, Stable; Coronary Artery Disease; Angina Pectoris, Variant; Ischemia; Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients and clinicians responsible for downstream (post-catheter laboratory) care are blinded to the randomisation allocation group (i.e. are blinded to whether the patient was in the intervention or blinded/control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Stratified Medicine (Active Comparator): All randomised participants will receive stratified medicine. The subjects will undergo functional coronary angiography involving guidewire-based coronary function tests (interventional diagnostic procedure, IDP) as an adjunct to invasive coronary angiography. The IDP results will be disclosed to the catheter laboratory clinician to clarify endotypes and re-evaluate the clinical diagnosis. Linked guideline-directed medical therapy and lifestyle measures will be recommended based on the endotype. The patient and clinicians responsible for downstream care will not be informed of the randomised group but they will be informed of the endotype and linked treatment plan, in the same way as in the Standard Care control group. They will be blinded to the allocated study arm and IDP findings.
  Interventions: Diagnostic Test: Disclosure of IDP results
- Standard Care Group (Sham Comparator): All randomised participants in this arm will receive standard angiography-guided care. The endotype will be determined based on the angiogram and all of the available clinical information. The participants in this group will also receive the IDP at time of the angiogram. The results of the IDP will be concealed from the catheter laboratory clinician who will be blinded. The cardiac physiologist / clinical scientist will remain unblinded for the purpose of data recording and quality assurance. The sham procedure is intended to be the same as in the Intervention Group. Management of the patient is as per standard of care, with therapy linked to the diagnosis (endotype). The patient and clinicians responsible for downstream care will not be informed of the randomised group but they will be informed of the endotype and linked treatment plan in the same way as in the Intervention Group. They will be blinded to the allocated study arm and IDP findings.
  Interventions: Other: IDP performed but results not disclosed

INTERVENTIONS:
Diagnostic Test: Disclosure of IDP results — The results of the adjunctive IDP performed at time of invasive coronary angiography are made available to the catheter laboratory clinician, to aid in the diagnostic process.
  Other Names: Stratified medicine
  Arms: Intervention Group - Stratified Medicine
Other: IDP performed but results not disclosed — The results of the IDP performed at the time of invasive coronary angiography are concealed from the catheter laboratory clinician who will be blinded. The patient is managed according to standard of care.
  Other Names: Standard, angiography-guided management
  Arms: Standard Care Group

SUMMARY:
The iCorMicA study is a multicentre, prospective, randomised, double-blind, sham-controlled, parallel-group, end-point trial and registry. The investigators seek to determine whether stratified medical therapy guided by an adjunctive interventional diagnostic procedure (IDP) during the invasive management of patients with known or suspected angina but no obstructive coronary artery disease improves symptoms, wellbeing, cardiovascular risk and clinical outcomes.

DETAILED DESCRIPTION:
Ischaemic heart disease (IHD) includes coronary artery disease (or 'coronary heart disease 'CHD') and ischaemic with no obstructive coronary arteries (INOCA). Coronary angiography is standard care for the evaluation of symptomatic patients and known or suspected coronary artery disease. A considerable proportion e.g. >1 in 3, of patients undergoing invasive coronary angiography for known or suspected angina do not have obstructive epicardial coronary artery disease.

The CorMicA pilot study involved prospective enrolment of patients referred for clinically indicated coronary angiography during a 12-month period (2016-2017) in the West of Scotland). 391 patients were enrolled, 185 (47%) had no obstructive coronary disease and 151 were randomised in a clinical trial of stratified medicine based on invasive tests of coronary vascular function. A high proportion (~4 in 5) of these patients had a diagnosis of INOCA due to a disorder of coronary vasomotion including microvascular- and/or vasospastic angina. The trial provided preliminary evidence that stratified medicine, as an adjunct to standard angiography-guided management, has potential to improve symptoms and quality of life. The mechanisms involved changes in diagnosis, treatment and lifestyle measures.

The CorMicA investigators were the first group to introduce stratified medicine for the management of ischaemic heart disease. Limitations of the CorMicA study included the setting (mainly single centre), partial blinding, short-term follow-up (primary outcome at 6 months) and the sample size. Acetylcholine reactivity testing was used to assess the susceptibility to coronary spasm (microvascular and/or macrovascular). Although acetylcholine is a naturally occurring substance, current formulations are not licensed for parenteral administration. Further, clinicians should have training and experience before implementing acetylcholine coronary reactivity testing. These considerations present a barrier to adoption in daily practice, which becomes all the more relevant given INOCA is generally under-recognised. A diagnostic coronary guidewire is already widely used in standard care and, unlike reactivity testing using acetylcholine, a guidewire has transferable potential to support stratified medicine during routine practice. This is especially the case for ad-hoc follow-on testing when obstructive coronary artery disease is excluded.

The vasoactive responses to acetylcholine reflect endothelial and vascular smooth muscle cell effects, which may overlap with the vasoactive responses to adenosine (non-endothelial dependent). Calcium channel blocker therapy is indicated for the functional endotypes associated with impaired vasodilatation and/or vasoconstriction. This raises the possibility that acetylcholine testing may not be routinely required as an adjunctive test to coronary angiography and instead could be reserved for selected cases, or in specialist centres. Instead, the diagnostic guidewire approach may be sufficient as a routine, first line test for the evaluation of INOCA during daily practice.

Anatomical imaging using coronary angiography is the standard of care and clinicians may determine any diagnosis based on all of the available information and their clinical judgement. This approach avoids the need for additional tests. With this approach, the patient's symptoms in response to empirical therapy can be assessed during follow-up and the treatment can be revised as clinically appropriate. In daily practice, adoption of adjunctive tests of coronary function is very low and, in the absence of large, multicentre trials, coronary angiography with or without adjunctive tests of coronary vascular function may be considered reasonable, reflecting equipoise.

iCorMicA is a multicentre, prospective, randomised, double-blind, sham-controlled, parallel-group, end-point (patient reported outcome measures (PROMS), health outcomes, health economics) trial and registry. The investigators aim to determine whether stratified medical therapy, guided by a guidewire-based interventional diagnostic procedure (IDP) at the time of invasive coronary angiography (i.e. functional angiography), improves outcomes in patients with known or suspected angina but no obstructive coronary artery disease. Symptoms of angina or angina-equivalent are determined according to the Rose and/or Seattle Angina questionnaires. The IDP utilises principles of thermodilution to measure coronary vascular function (IMR, CFR, RRR), which aid clinicians in establishing a diagnosis of microvascular angina, vasospastic angina, mixed (both), or none, as per Coronary Vasomotion Disorders International Study Group (COVADIS) criteria. The feasibility, safety, efficacy and effect on healthcare resource utilisation of stratified medicine will be tested in multiple hospitals in different countries in Europe.

Participants with no obstructive epicardial coronary artery disease (coronary stenosis <50% and/or FFR >0.80) are eligible for randomisation (1:1) to either the intervention (IDP-guided, results disclosed) or blinded control (IDP undertaken but results not disclosed, standard of care) group. Medical therapy will be informed according to the clinical diagnosis (endotype). Patients in the intervention group with abnormal coronary vascular function may undergo repeated evaluations to assess the response to intracoronary therapy e.g. calcium channel blocker, enabling a personalised treatment plan. Patients who are ineligible for randomisation (e.g. obstructive coronary artery disease) may be entered into a prospective clinical registry, with individuals from each site invited to undergo similar follow-up assessments as the randomised participants.

Trial participants will be blinded to treatment group. The clinicians responsible for on-going care will also be blinded. Following invasive management, patients and clinicians will be advised of the diagnosis (endotype) but not the randomised group. The endotype will be informed by the IDP in the intervention group but not in the control group (sham procedure). Medical therapy and lifestyle measures are linked to the endotype and informed by contemporary practice guidelines. Therefore, optimal guideline-directed medical care according to the endotype is intended to be the same, regardless of the group allocation.

The sample size is 1500 randomised participants. The minimum follow-up duration is 12 months from the last participant recruitment. Follow-up will continued in the longer term including, where feasible, electronic case record linkage. The primary outcome measure is the Summary Score of the Seattle Angina Questionnaire at 12 months. Secondary outcomes include other Patient Reported Outcome Measures (PROMS) to describe other aspects of health and wellbeing. These include EQ-5D-5L, Illness perception (Brief IPQ), Treatment satisfaction (TSQM), Duke Activity Status Index (DASI), the International Physical Activity Questionnaire (IPAQ-SF) short-form and a pain questionnaire.

Additional objectives include the wider evaluation of the safety and diagnostic utility of the IDP in a multicentre, multinational setting, and the effects of stratified medicine on the rates of major adverse cardiovascular events by randomised group. The registry will represent a parallel control group. Scientific analyses of circulating biomarkers will be performed to better understand the pathophysiology of INOCA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. A clinical plan for invasive coronary angiography.
3. Symptoms of angina (typical or atypical) according to the Rose- and/or Seattle Angina questionnaires.
4. Able to comply with study procedures.
5. Able to provide informed consent.

Exclusion Criteria:

1. A non-coronary primary indication for invasive angiography (e.g. valve disease, heart failure).
2. History of coronary artery bypass surgery.
3. Presence of obstructive disease evident in a main coronary artery (diameter >2.5 mm), i.e. a coronary stenosis >50% and/or a fractional flow reserve (FFR) ≤0.80*.
4. Logistical reason*. *These patients will enter a follow-up registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire (SAQ) Summary Score | 12 months
  The 7-item version of the SAQ reflects the frequency of angina (SAQ Angina Frequency score) and the disease-specific effect of angina on patients' physical function (SAQ Physical Limitation score) and quality of life (Quality of Life score) over the previous 4 weeks; these scores are averaged to obtain the SAQ Summary score, which is an overall measure of patients' stable ischaemic heart disease-specific health status. SAQ scores range from 0 to 100, with higher scores indicating less frequent angina, improved function, and better quality of life.

SECONDARY OUTCOMES:
Feasibility of stratified medicine | 0-60 months
  Rates of enrolment, drop-out, completion of diagnostic protocol, integrity of blinding in the catheter laboratory and blinding at 1 year, loss to follow-up.
Safety of the interventional diagnostic procedure (IDP) | 0-60 months
  As reflected by SAEs related to the procedure, and those arising during longer term follow-up.
Diagnostic utility of the interventional diagnostic procedure (IDP) | 0-60 months
  To assess impact of disclosure of the coronary function test results on the diagnosis and certainty of the diagnosis. A missed diagnosis of microvascular angina is defined as a physician diagnosis of non-cardiac chest pain in the presence of objective abnormalities of coronary artery function.
Clinical utility | 0-60 months
  To assess the impact of disclosure of coronary function test results on clinical management (including treatment medication, investigations and healthcare resource utilisation).
Health status | 0-60 months
  To assess quality of life, symptoms and health status using validated, patient-administered questionnaires. The EQ5D, SAQ, angina diary, EQ-5D-5L, Brief IPQ, TSQM, DASI, IPAQ-SF, FSQ and MOCA questionnaires will be completed.
Cardiovascular risk | 0-60 months
  To assess attainment of guideline targets for measured cardiovascular risk factors, and adherence.
Health outcomes | 0 months - 10 years
  MACE including death, re-hospitalisation for cardiovascular events including myocardial infarction, heart failure, stroke/ TIA, unstable angina and coronary revascularisation. Unscheduled hospital visits for chest pain that have not led to hospital admission will also be documented.
Health economics | 0 months - 10 years
  Health resource utilisation will also be assessed by identifying inpatient visits, procedures and medication use.

OTHER OUTCOMES:
Cardiovascular biomarkers | 0 months - 10 years
  Hypothesis: Compared with standard care, stratified medicine improves circulating biomarkers of cardiovascular risk
Sex differences | 0 months - 10 years
  To assess for similarities and differences in presenting characteristics, socio-economic status, treatment, health status and clinical outcomes between males and females.
Ischaemic heart disease | 0 months - 10 years
  To assess for similarities and differences in presenting characteristics, socio-economic status, treatment, health status and clinical outcomes between patient with obstructive coronary artery disease and no obstructive CAD (including by endotype).

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, MBChB, PhD, Study Chair — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Golden Jubilee National Hospital, Clydebank, Scotland
  - NHS Greater Glasgow and Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the study has completed
Access Criteria: Bone fide collaboration request
URL: http://www.gla.ac.uk/researchinstitutes/icams/staff/colinberry/

REFERENCES:
- [Background] Kunadian V, Chieffo A, Camici PG, Berry C, Escaned J, Maas AHEM, Prescott E, Karam N, Appelman Y, Fraccaro C, Louise Buchanan G, Manzo-Silberman S, Al-Lamee R, Regar E, Lansky A, Abbott JD, Badimon L, Duncker DJ, Mehran R, Capodanno D, Baumbach A. An EAPCI Expert Consensus Document on Ischaemia with Non-Obstructive Coronary Arteries in Collaboration with European Society of Cardiology Working Group on Coronary Pathophysiology & Microcirculation Endorsed by Coronary Vasomotor Disorders International Study Group. Eur Heart J. 2020 Oct 1;41(37):3504-3520. doi: 10.1093/eurheartj/ehaa503. PMID 32626906
- [Background] Bairey Merz CN, Pepine CJ, Walsh MN, Fleg JL. Ischemia and No Obstructive Coronary Artery Disease (INOCA): Developing Evidence-Based Therapies and Research Agenda for the Next Decade. Circulation. 2017 Mar 14;135(11):1075-1092. doi: 10.1161/CIRCULATIONAHA.116.024534. PMID 28289007
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] Jespersen L, Hvelplund A, Abildstrom SZ, Pedersen F, Galatius S, Madsen JK, Jorgensen E, Kelbaek H, Prescott E. Stable angina pectoris with no obstructive coronary artery disease is associated with increased risks of major adverse cardiovascular events. Eur Heart J. 2012 Mar;33(6):734-44. doi: 10.1093/eurheartj/ehr331. Epub 2011 Sep 11. PMID 21911339
- [Background] Sara JD, Widmer RJ, Matsuzawa Y, Lennon RJ, Lerman LO, Lerman A. Prevalence of Coronary Microvascular Dysfunction Among Patients With Chest Pain and Nonobstructive Coronary Artery Disease. JACC Cardiovasc Interv. 2015 Sep;8(11):1445-1453. doi: 10.1016/j.jcin.2015.06.017. PMID 26404197
- [Background] Ford TJ, Yii E, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, McCartney P, Corcoran D, Collison D, Rush C, Stanley B, McConnachie A, Sattar N, Touyz RM, Oldroyd KG, Berry C. Ischemia and No Obstructive Coronary Artery Disease: Prevalence and Correlates of Coronary Vasomotion Disorders. Circ Cardiovasc Interv. 2019 Dec;12(12):e008126. doi: 10.1161/CIRCINTERVENTIONS.119.008126. Epub 2019 Dec 13. PMID 31833416
- [Background] Ford TJ, Stanley B, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, McCartney P, Corcoran D, Collison D, Rush C, Sattar N, McConnachie A, Touyz RM, Oldroyd KG, Berry C. 1-Year Outcomes of Angina Management Guided by Invasive Coronary Function Testing (CorMicA). JACC Cardiovasc Interv. 2020 Jan 13;13(1):33-45. doi: 10.1016/j.jcin.2019.11.001. Epub 2019 Nov 11. PMID 31709984
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Ong P, Camici PG, Beltrame JF, Crea F, Shimokawa H, Sechtem U, Kaski JC, Bairey Merz CN; Coronary Vasomotion Disorders International Study Group (COVADIS). International standardization of diagnostic criteria for microvascular angina. Int J Cardiol. 2018 Jan 1;250:16-20. doi: 10.1016/j.ijcard.2017.08.068. Epub 2017 Sep 8. PMID 29031990
- [Derived] Ang DTY, Collison DG, McGeoch RJ, Carrick D, Sykes RA, Bradley C, Kamdar AL, Jong A, Brogan RA, MacDougall DA, McCartney PJ, Rocchiccioli JP, Apps AP, Murphy CA, Robertson KE, Shaukat A, Ghattas A, Joshi FR, Sood A, Good RIS, O'Rourke B, Eteiba H, Lindsay MM, McConnachie A, Berry C. Novel Contrast-Derived Indices of Coronary Microvascular Function: Potential Clinical and Cost Benefits. Circ Cardiovasc Interv. 2025 Jun;18(6):e015058. doi: 10.1161/CIRCINTERVENTIONS.124.015058. Epub 2025 May 1. PMID 40308206